CLINICAL TRIAL: NCT03656770
Title: Measuring Beliefs and Norms About Persons With Mental Illness in Rural Uganda: A Randomized Survey Experiment
Brief Title: Measuring Beliefs and Norms About Persons With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Alexander Tsai, Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2013P000395
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Mental Illness; Schizophrenia; Bipolar Disorder; Depression
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Bipolar Disorder; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- V1: Control (No Intervention): This version of the survey questionnaire depicts a young woman with no symptoms of mental illness.
- V2: Schizophrenia (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with untreated and symptomatic schizophrenia.
  Interventions: Other: Survey questionnaire
- V3: Schizophrenia + Tx with Response (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with schizophrenia, successfully treated with complete response.
  Interventions: Other: Survey questionnaire
- V4: Schizophrenia + Tx with Relapse (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with schizophrenia, successfully treated with partial relapse.
  Interventions: Other: Survey questionnaire
- Version 5: Bipolar (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with untreated and symptomatic bipolar disorder.
  Interventions: Other: Survey questionnaire
- V6: Bipolar + Tx with Response (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with bipolar disorder, successfully treated with complete response.
  Interventions: Other: Survey questionnaire
- V7: Bipolar + Tx with Relapse (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with bipolar disorder, successfully treated with partial relapse.
  Interventions: Other: Survey questionnaire
- V8: Depression (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with untreated and symptomatic major depressive disorder.
  Interventions: Other: Survey questionnaire
- V9: Depression + Tx with Response (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with major depressive disorder, successfully treated with complete response.
  Interventions: Other: Survey questionnaire
- V10: Depression + Tx with Relapse (Experimental): As this is a survey experiment, the "intervention" involves random assignment to a survey questionnaire with specific wording. This version of the survey questionnaire depicts a young woman with major depressive disorder, successfully treated with partial relapse.
  Interventions: Other: Survey questionnaire

INTERVENTIONS:
Other: Survey questionnaire — Each version of the questionnaire portrays a young Ugandan woman with different profiles of illness severity, treatment, and treatment response.
  Arms: V10: Depression + Tx with Relapse; V2: Schizophrenia; V3: Schizophrenia + Tx with Response; V4: Schizophrenia + Tx with Relapse; V6: Bipolar + Tx with Response; V7: Bipolar + Tx with Relapse; V8: Depression; V9: Depression + Tx with Response; Version 5: Bipolar

SUMMARY:
Survey experiment to estimate drivers of mental illness stigma

DETAILED DESCRIPTION:
Despite significant advances in scientific understanding of brain and substance use disorders accompanied by significant advances in treatment and improvements in prognosis, mental illness remains highly stigmatized throughout the world. Previous studies suggest that portraying mental illness as treatable can reduce negative attitudes toward persons with mental illness. This randomized controlled trial compares the effects of exposing study participants to vignettes portraying persons with untreated and symptomatic mental illness vs. treated mental illness with complete response vs. treated mental illness with relapse. It is hypothesized, based on prior work, that study participants exposed to vignettes depicting treated mental illness with completed response would have the greatest effect on reducing negative attitudes toward persons with mental illness, followed by treated mental illness with relapse and untreated and symptomatic mental illness.

ELIGIBILITY:
Inclusion Criteria:

* all persons who considered Nyakabare Parish their primary place of residence and who were capable of providing consent

Exclusion Criteria:

* minors younger than 18 years of age, with the exception of emancipated minors
* persons who did not consider Nyakabare their primary place of residence, e.g., persons who happened to be visiting Nyakabare at the time of the survey or who owned a home in Nyakabare but spent most of their time outside the parish
* persons with whom research staff could not communicate, e.g., due to deafness, mutism, or aphasia
* persons with psychosis, neurological damage, acute intoxication, or other cognitive impairment (all of which were determined informally in the field by non-clinical research staff in consultation with a supervisor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1782 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

PRIMARY OUTCOMES:
Social Distance | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Willingness to have the woman portrayed in the vignette to marry into the study participant's family (single item culturally adapted instrument developed specifically for this study)
Perceived Norms about Social Distance | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Study participant's perception of the extent to which other people would be willing to have the woman portrayed in the vignette to marry into their families (single item culturally adapted instrument developed specifically for this study)
Negative Attitudes (Attribution) | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Personal belief that the symptoms of the woman portrayed in the vignette represent divine punishment (single item culturally adapted instrument developed specifically for this study)
Perceived Norms about Negative Attitudes (Attribution) | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Study participant's perception of the extent to which other people believe that the symptoms of the woman portrayed in the vignette represent divine punishment (single item culturally adapted instrument developed specifically for this study)
Negative Attitudes (Shame) | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Personal belief that the symptoms of the woman portrayed in the vignette bring shame upon her family
Perceived Norms about Negative Attitudes (Shame) | Immediate (assessed with respect to the study participant's beliefs at a single time point, which is the time at which the survey is administered)
  Study participant's perception of the extent to which other people believe that the symptoms of the woman portrayed in the vignette bring shame upon her family (single item culturally adapted instrument developed specifically for this study)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander C Tsai, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rasmussen JD, Kakuhikire B, Baguma C, Ashaba S, Cooper-Vince CE, Perkins JM, Bangsberg DR, Tsai AC. Portrayals of mental illness, treatment, and relapse and their effects on the stigma of mental illness: Population-based, randomized survey experiment in rural Uganda. PLoS Med. 2019 Sep 20;16(9):e1002908. doi: 10.1371/journal.pmed.1002908. eCollection 2019 Sep. PMID 31539373